CLINICAL TRIAL: NCT03925987
Title: Predicting Treatment Response to Exposure Therapy Using a CO2 Habituation Paradigm in Patients With High Levels of Anxiety Sensitivity
Brief Title: Predicting Treatment Response to Exposure Therapy Using Carbon Dioxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CoBRE CO2
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Agoraphobia
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Agoraphobia | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure therapy (Experimental): Participants complete 10 weekly sessions of a group-based exposure therapy class for anxiety disorders.
  Interventions: Behavioral: Exposure therapy

INTERVENTIONS:
Behavioral: Exposure therapy — 10 weekly sessions of group-based exposure therapy

SUMMARY:
Anxiety disorders affect over a quarter of the population, yet very little is known about the variables that predict treatment outcome. The planned study explores whether a patient's response to a physiological test involving inhalation of carbon dioxide predicts their response to exposure therapy.

DETAILED DESCRIPTION:
Anxiety Sensitivity (AS) refers to an individual's fear of experiencing anxiety-related symptoms (e.g., dyspnea or heart palpitations) and is a core construct underlying the initiation and maintenance of pathological anxiety. Recent evidence suggests that reducing AS may be critical for the prevention and treatment of anxiety across diagnostic categories. Exposure therapy, an important component of cognitive behavioral therapy (CBT), is one of the most effective treatments for reducing AS, and has been shown to improve symptoms across a number of different anxiety disorders. Meta-analyses reveal an approximately 50% treatment response rate, with the remaining half of patients showing either no response or dropping out of treatment early. Unfortunately, there is a paucity of research exploring which variables predict treatment outcome and there are currently no tests for predicting which patients would benefit the most from exposure therapy. In this study, participants will complete two sessions of a carbon dioxide (CO2) habituation paradigm, a safe and noninvasive physiological test that entails repeated exposures to single vital capacity inhalations of 20% CO2. Both CO2 testing sessions will be completed within a 72-hour time period. Patients then complete a 10-week group-based exposure therapy to determine whether an individual's degree of habituation to CO2 predicts treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-V diagnosis of an Anxiety disorder (Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia)
2. Anxiety Sensitivity Index (ASI-3) total score > 29
3. Overall Anxiety Severity and Impairment Scale (OASIS) score > 8
4. Between 18-55 years of age
5. Subject must be "treatment-seeking" and willing to enroll in the 10-week group-based Exposure Therapy

Exclusion Criteria:

1. Comorbid Bipolar Disorder, Schizophrenia, Anorexia or Bulimia Nervosa, or Obsessive-Compulsive Disorder
2. Current Substance Use Disorder > moderate (within the past 6 months)
3. Currently taking a psychotropic medication
4. Currently receiving psychotherapy/counseling for anxiety
5. Currently being treated as an inpatient
6. Active suicidal ideation with intent or plan
7. History of neurological, cardiovascular or respiratory problems (e.g., asthma, severe brain injury)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Between-session habituation of self-reported anxiety | Across two days of CO2 testing within a 72-hour window
  Maximum anxiety rating on a 10-point rating dial (0=no anxiety to 10=most anxiety ever) during day 1 of CO2 testing minus the maximum anxiety rating during day 2 of CO2 testing

SECONDARY OUTCOMES:
Between-session habituation of self-reported dyspnea | Across two days of CO2 testing within a 72-hour window
  Dyspnea rating (difficulty breathing, shortness of breath or smothering) on a 100-point visual analogue scale (0=not at all to 100=extremely) during day 1 of CO2 testing minus the dyspnea rating during day 2 of CO2 testing
Between-session reduction in avoidance behavior | Across two days of CO2 testing within a 72-hour window
  Average response latency (in seconds) between vital capacity breaths of CO2 during day 1 of CO2 testing minus the average response latency during day 2 of CO2 testing

CONTACTS AND LOCATIONS:
Overall Officials: Justin Feinstein, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03925987/ICF_000.pdf